CLINICAL TRIAL: NCT05359887
Title: PET-study on the Role of the Reward System in Weight Loss After Bariatric Surgery
Acronym: ObesiPET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UMCG202100632
Record Dates: First submitted 2022-04-12; First posted 2022-05-04 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Obesity
Keywords: Obesity; Reward system; PET-scan; [11C]-Raclopride
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unsuccessful BS (Total Weight Loss (TWL) < 20%) (Experimental): Fifteen who had unsuccessful BS (Total Weight Loss (TWL) < 20%)
  Interventions: Other: standardized liquid mixed meal Nutridrink®
- Successful BS (TWL > 25%). (Experimental): Fifteen who had successful BS (TWL > 25%).
  Interventions: Other: standardized liquid mixed meal Nutridrink®

INTERVENTIONS:
Other: standardized liquid mixed meal Nutridrink® — Administration of food in controlled situation

SUMMARY:
Bariatric surgery (BS) is currently the most effective treatment in severe obesity. However, a considerable percentage of patients undergoing BS fail to lose sufficient weight or regain weight after initial weight loss during long-term follow-up, which may be attributed to personality traits and pathological eating behaviour. Previous positron emission tomography (PET) studies have shown reduced dopamine D2 receptor availability in obese patients and upregulation of this availability following successful BS in the brain's reward system. Dopamine D2 receptor availability in patients with unsuccessful BS has not been investigated to date.

ELIGIBILITY:
Inclusion Criteria:

* Bariatric surgery 24-36 months prior to the study
* Adult (over 18y old)
* Mentally capable to understand the consequences of the procedure and make his or her own choice without coercion
* Able to undergo PET and MRI, according to the investigator's assessment
* Native speaking
* Able to participate in follow-up
* Written informed consent

Exclusion Criteria:

* Presence of a DSM-IV axis 1 disorder
* The use of drugs that bind to dopamine D2/3 receptors, including various classes of antipsychotics and antidepressants
* History of stroke, brain tumor, Parkinson's Disease or dementia
* History of head trauma with loss of consciousness
* Alcohol or substance abuse in the last 6 months
* Alcohol consumption 24h prior to PET scanning
* Smoking or other forms of nicotine intake 12 hours prior to PET scanning
* Use of anorectic drugs in the last 6 months
* Current pregnancy
* Medication for Diabetes Mellitus
* Claustrophobia
* The presence of implanted metal objects of the type which may concentrate radiofrequency fields or cause tissue damage from twisting in a magnetic field (such as certain implanted devices, shrapnel, ocular metal shavings)
* Patients with a bodyweight > 200kg will be excluded to ensure the maximum load of the camera bed of the PET-scanner (227 kg) is not exceeded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in [11C]-raclopride binding potential in the brain's reward system between study groups before and after a food challenge. | -50 minutes (before start of PET scanning), 0 minutes (during PET break, before mixed meal), 30 minutes (after second phase of PET-scanning)
  Pre- and post-eating changes in dopamine D2 receptor availability as indexed by the [11C]-raclopride binding potential in the brain's reward system between subjects who underwent successful vs unsuccessful bariatric surgery

SECONDARY OUTCOMES:
The correlation between [11C]-raclopride binding potential in the brain's reward system and of questionnaires and diaries | Pre-intervention
  The correlation between questionnaires on eating habits (EDE-Q, REO, YFAS) and quality of life (OBESI-Q) in patients who had successful vs unsuccessful BS and [11C]-raclopride binding potential.
The correlation between [11C]-raclopride binding potential in the brain's reward system and of gut hormones. | -50 minutes (before start of PET scanning), 0 minutes (during PET break, before mixed meal), 30 minutes (after second phase of PET-scanning), 60 - 90 - 120 minutes
  The relation between fasting or fed (gut) hormone concentrations and dopamine D2 receptor availability in the reward system.

CONTACTS AND LOCATIONS:
Locations (1):
- MCL, Leeuwarden, Netherlands

IPD SHARING:
Plan to Share IPD: No